CLINICAL TRIAL: NCT02202473
Title: Oxymatrine Plus Lamivudine Combination Therapy Versus Lamivudine Monotherapy for Chronic Hepatitis B Infected Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Southeast University, China (Other)
Collaborators: Cttq (Industry)
Responsible Party: Principal Investigator, Wei Zhao, director of the hospital, Southeast University, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Oxymatrine
Record Dates: First submitted 2014-07-24; First posted 2014-07-29 (Estimated); Last update posted 2014-07-29 (Estimated); Status verified 2014-07

CONDITIONS: Chronic Hepatitis B
Keywords: Oxymatrine Capsules, lamivudine, chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Lamivudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lamivudine (Active Comparator): Lamivudine (Manufacturer: GlaxoSmithKline) 100mg po, qd
  Interventions: Drug: Lamivudine
- Lamivudine+Oxymatrine Capsules (Experimental): Lamivudine (Manufacturer: GlaxoSmithKline) 100mg po, qd; oxymatrine Capsules (Chia Tai Tianqing Pharmaceutical Group Co., Ltd) 200 mg, po, tid.
  Interventions: Drug: Lamivudine+Oxymatrine Capsules

INTERVENTIONS:
Drug: Lamivudine
  Arms: Lamivudine
Drug: Lamivudine+Oxymatrine Capsules
  Arms: Lamivudine+Oxymatrine Capsules

SUMMARY:
The purpose of this study is to evaluate the efficacy of Oxymatrine plus Lamivudine Combination Therapy and whether it could lower the incidence of Lamivudine long-term resistance compared to Lamivudine Monotherapy.

DETAILED DESCRIPTION:
Group A (Lamivudine Monotherapy): Lamivudine (Manufacturer: GlaxoSmithKline) 100mg po, qd.

Group B (Oxymatrine + Lamivudine Combination Therapy): Lamivudine (Manufacturer: GlaxoSmithKline) 100mg po, qd; oxymatrine Capsules (Chia Tai Tianqing Pharmaceutical Group Co., Ltd) 200 mg, po, tid.

Total subjects: 200, 100 patients randomized in each group.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 60 years old.
2. Subjects diagnosed as chronic hepatitis B according to 2000 Xi'an Conference Guidelines: Management of chronic hepatitis B. Alanine transaminase >80 IU/L, total bilirubin<85.5 mmol/L, Hepatitis B virus DNA >1×10^5copies/mL; haven't been treated with antiviral therapy within 6 months before screening.
3. able to give written informed consent and to comply with the study protocol.
4. Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study.

Exclusion Criteria:

1. Evidence of hepatocellular carcinoma
2. Clinical symptoms of Decompensated liver disease at screening, including but not limited to: Serum bilirubin≥1.5 x upper limit of normal, prothrombin time of greater than 2 seconds prolonged, a serum albumin< 32g/L, or a history of ascites, variceal bleeding, or hepatic encephalopathy;
3. Alanine transaminase>10 x upper limit of normal at screening or history of Transient hepatic decompensation caused by acute exacerbation;
4. hemoglobin< 10g/dL, Neutrophil count<1.5 × 10^9/L, platelet count< 80 × 10^9/L;
5. Evidence of active liver disease from other causes, including co-infection with hepatitis A virus, co-infection with hepatitis E virus, co-infection with hepatitis C virus, co-infection with hepatitis D virus, co-infection with HIV, autoimmune hepatitis (antinuclear antibody titer> 1:100);
6. Use of immunosuppressors, immunomodulators (including interferon or thymosin) within 6 months before enrollment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 192 (Actual)
Dates: Primary Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Reduction of Hepatitis B virus DNA titer compared to Baseline Hepatitis B virus DNA titer every 3 months for 18 months | 1, 3, 6, 12, 15, 18 months

SECONDARY OUTCOMES:
Hepatitis B virus resistance loci | 1, 3, 6, 12, 15, 18 months

CONTACTS AND LOCATIONS:
Locations (1):
- the second hospital of Nanjing, Nanjing, Jiangsu, China

REFERENCES:
- [Background] Lu FM, Zhuang H. Management of hepatitis B in China. Chin Med J (Engl). 2009 Jan 5;122(1):3-4. No abstract available. PMID 19187608
- [Background] Yuen MF, Fung J, Wong DK, Lai CL. Prevention and management of drug resistance for antihepatitis B treatment. Lancet Infect Dis. 2009 Apr;9(4):256-64. doi: 10.1016/S1473-3099(09)70056-8. PMID 19324298
- [Background] Wang YP, Zhao W, Xue R, Zhou ZX, Liu F, Han YX, Ren G, Peng ZG, Cen S, Chen HS, Li YH, Jiang JD. Oxymatrine inhibits hepatitis B infection with an advantage of overcoming drug-resistance. Antiviral Res. 2011 Mar;89(3):227-31. doi: 10.1016/j.antiviral.2011.01.005. Epub 2011 Jan 28. PMID 21277330